CLINICAL TRIAL: NCT04097418
Title: Effects of Aerobic Training on Motor and Cognitive Performances in Patients With MS: an Exploratory Study With Structural and Functional MRI
Brief Title: Aerobic Training Effects on Motor and Cognitive Performances in MS: an Exploratory Study With Structural and Functional MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Prof. Massimo Filippi, Head of Neurology, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Training aerobico-SM 2015
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Aerobic Training; rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: This study is a monocentric, non-pharmacological, longitudinal, randomized, blind, controlled study.
  Subjects The Investigators will study 40 MS patients and 40 HC. Subjects will then be randomized through a sequence generated by the computer to determine their assignment to the conventional motor rehabilitation therapy group (control group) or to the aerobic training (experimental group). The computerized randomization software will generate personal codes to allocate every patient to a treatment arm.
  Participants will be split into 4 groups of 20 subjects per group:
  1. Group of aerobic training of healthy subjects: aerobic training by treadmill at moderate intensity;
  2. Group of conventional motor training of healthy subjects: training of passive mobility, stretching and balance;
  3. Group of aerobic training of MS patients: aerobic training by treadmill at moderate intensity;
  4. Treatment group control of MS patients: training of passive mobility, stretching and balance.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The computerized randomization software will generate personal codes to allocate every patient to a treatment arm. These codes will be placed in opaque envelopes and delivered to the patient by an operator external to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aerobic training in healthy subjects (Experimental): For each healthy subject, the treatment will lasts 8 weeks. Each treatment will consists of 35 minutes of training, administered 3 times per week.
  Subjects of the experimental groups (both patients and healthy controls) will carry out an aerobic training of moderate intensity (fixed time and variable intensity) on a treadmill. The training will be set individually via direct method: during the first session, the subject will be trained at an intensity that gets the heart rate (HR) corresponding to 46-63% of VO2 peak measured during the exercise test; in subsequent sessions the intensity will increase to maintain the same HR, which will be always monitored. The intensity workout identified will be maintained for 30 minutes each session, preceded and followed by a few minutes of warm-up and cool-down.
  Interventions: Behavioral: Aerobic training compared to conventional motor training
- Conventional motor training of healthy subjects (Active Comparator): For each healthy subject, the treatment will lasts 8 weeks. Each treatment will consists of 35 minutes of training, administered 3 times per week.
  Control groups of both patients and healthy subjects will follow a conventional non-aerobic physiotherapy training, structured in: 15 minutes of passive mobilization of upper and lower limbs and spine, 5 minutes of stretching of the upper and the lower limbs and 10 minutes of balance training.
  Interventions: Behavioral: Aerobic training compared to conventional motor training
- Aerobic training in MS patients (Experimental): For each MS patient, the treatment will lasts 8 weeks. Each treatment will consists of 35 minutes of training, administered 3 times per week.
  Subjects of the experimental groups (both patients and healthy controls) will carry out an aerobic training of moderate intensity (fixed time and variable intensity) on a treadmill. The training will be set individually via direct method: during the first session, the subject will be trained at an intensity that gets the heart rate (HR) corresponding to 46-63% of VO2 peak measured during the exercise test; in subsequent sessions the intensity will increase to maintain the same HR, which will be always monitored. The intensity workout identified will be maintained for 30 minutes each session, preceded and followed by a few minutes of warm-up and cool-down.
  Interventions: Behavioral: Aerobic training compared to conventional motor training
- Conventional motor training of MS patients (Active Comparator): For each MS patient, the treatment will lasts 8 weeks. Each treatment will consists of 35 minutes of training, administered 3 times per week.
  Control groups of both patients and healthy subjects will follow a conventional non-aerobic physiotherapy training, structured in: 15 minutes of passive mobilization of upper and lower limbs and spine, 5 minutes of stretching of the upper and the lower limbs and 10 minutes of balance training.
  Interventions: Behavioral: Aerobic training compared to conventional motor training

INTERVENTIONS:
Behavioral: Aerobic training compared to conventional motor training — Aerobic training: aerobic training by treadmill at moderate intensity. Each treatment will consists of 35 minutes of training, administered 3 times per week, for 8 weeks.
  Conventional motor training: 15 minutes of passive mobilization of upper and lower limbs and spine, 5 minutes of stretching of the upper and the lower limbs and 10 minutes of balance training, administered 3 times per week, for 8 weeks.
  Other Names: Conventional motor training

SUMMARY:
Aerobic training (AT) induces cardiovascular, metabolic and muscular changes and has been proposed as a promising rehabilitative approach in elderly adults and in neurological patients to improve both motor and cognitive performances. The Investigators wish to explore the role of AT in multiple sclerosis (MS) patients on physical and neuropsychological functions and its underlying anatomical and functional substrates, using advanced magnetic resonance imaging (MRI) methods.

In this project, the Investigators wish to apply aerobic training in right-handed MS patients and healthy controls to assess:

1. the effects of aerobic training compared to conventional motor training on motor and cardio-vascular parameters;
2. the effect of aerobic training compared to conventional motor training on cognitive performance, depression and fatigue;
3. the modifications of functional activations during a cognitive task and of functional connectivity in motor and cognitive networks during resting state following aerobic training and conventional motor training (functional plasticity);
4. the regional variations of gray matter (GM) volumes and white matter (WM) architecture after aerobic training and conventional motor training (structural plasticity);
5. the correlations between the changes detected with structural and functional MRI and clinical, motor and neuropsychological scales.

DETAILED DESCRIPTION:
This study is a monocentric, non-pharmacological, longitudinal, randomized, blind, controlled study.

Subjects The Investigators will study 40 right-handed MS patients with Expanded Disability Status Scale (EDSS) score ≤6 and an indication to perform a physiotherapy treatment by the treating physician. Patients will be recruited from the Department of Neurology, San Raffaele Hospital. Forty sex- and age-matched right-handed healthy individuals (HC) will also be enrolled. The HC will be recruited from the patients' relatives or acquaintances of the study personnel. The enrolment of HC is crucial to define whether post-treatment changes observed in MS patients are adaptive or maladaptive and to estimate the magnitude of these alterations.

Subjects who will satisfy the inclusion criteria will then be randomized through a sequence generated by the computer to determine their assignment to the conventional motor rehabilitation therapy group (control group) or to the aerobic training (experimental group). The computerized randomization software will generate personal codes to allocate every patient to a treatment arm. These codes will be placed in opaque envelopes and delivered to the patient by an operator external to the study.

Thus, participants will be split into 4 groups of 20 subjects per group:

1. Experimental group of HC: aerobic training by treadmill at moderate intensity;
2. Control group of HC: training of passive mobility, stretching and balance;
3. Experimental group of MS patients: aerobic training by treadmill at moderate intensity;
4. Control group of MS patients: training of passive mobility, stretching and balance.

   Inclusion criteria (All)
   * Age: 18-65 years;
   * Native italian language speaking;
   * Right-handed;
   * No particular motor skills;
   * No additional neurologic, psychiatric, orthopaedic or rheumatologic diseases;
   * Normal or corrected-to-normal vision;
   * No MRI contraindications;
   * Ability to understand the purpose of the study and provide signed informed consent.

   For MS patients, the following additional inclusion criteria will be applied:
   * Patients with a MS diagnosis;
   * EDSS ≤6.0;
   * Stable MS treatment from ≥1 month prior to study enrolment;
   * Relapse- and steroid-free from ≥3 months before screening visit;
   * An indication to perform a physiotherapy treatment by the treating physician.

   Exclusion criteria
   * Persons who perform regularly a structured training;
   * Patients who performed a physiotherapy treatment for at least 3 months;
   * Concomitant therapy with antidepressant, baclofen, psychoactive, and steroids drugs as well as symptomatic treatment for fatigue;
   * History of alcohol or substance abuse;
   * Pregnancy or breastfeeding.

   Clinical and functional assessment All subjects will undergo a screening questionnaire and a cardiologic evaluation, including electrocardiogram, followed by a graded exercise test, in order to exclude possible contraindications to the inclusion in the study.

   The graded exercise test will permit to measure the following parameters:
   * peak oxygen consumption (VO2);
   * maximum wattage;
   * heart rate (isolabour and maximum);
   * rate of perceived exertion (Borg scale of rating of perceived exertion (RPE)).

   Subjects who will satisfy the inclusion criteria will be randomized to the four groups previously described.

   All the subject will be assessed with clinical, cardiologic, neuropsychological and MRI evaluations at:
   * baseline (before the start of the rehabilitation treatment) - T0,
   * Week 4 - T1,
   * Week 8 (end of the study) - T2. A clinical follow-up has been planned 3 months after the end of the treatment.

   At each time-point, MS patients will be evaluated with the following assessments:
   * Graded exercise test;
   * Complete neurological evaluation by a neurologist with the definition of the EDSS score and the MS Functional Composite (MSFC);
   * Assessment of autonomy in daily life activities, through the "Functional Independence Measurement" (FIM);
   * Spasticity, evaluating the modified Ashworth scale;
   * Fatigue, through the Modified Fatigue Impact Scale (MFIS);
   * Depression, using the Beck Depression Inventory II (BDI-II);
   * Perceived quality of life, through the Multiple Sclerosis Quality of Life Scale (MSQOL-54).

   HC will be evaluated with the MSFC, MFIS and BDI-II. All subjects will also be evaluated on additional motor aspects by the "6 minutes walking test" and the "Time up and go" test. Finally, participants will undergo a neuropsychological assessment, using the Brief Repeatable Battery of Neuropsychological Tests, the Digit Span (forward and backward) and the Brief Test of Intelligence.

   At the same time-points, all subjects will perform a MR scan, using a 3.0 Tesla scanner, available at the San Raffaele Hospital. The following brain MRI sequences will be acquired:
   1. Dual-echo (DE) turbo spin echo (SE);
   2. 3D T1-weighted fast field echo;
   3. Pulsed-SE gradient echo planar imaging (EPI) with SENSE (acceleration factor=2) and diffusion gradients applied in 35 non-collinear directions;
   4. functional MRI (fMRI) in Resting State (RS) condition;
   5. fMRI with an active cognitive task (Stroop task): using an event-related design, it will be proposed different type of stimuli, i.e. congruent, incongruent and neutral stimuli. Participants will be asked to respond to the color of the ink through four buttons (red, green, yellow, blue) of a fMRI compatible response-box, which will record reaction times and accuracy.

   Assessors of clinical, neuropsychological and MRI evaluations will be blind with respect to participants allocation.

   Safety Possible fatigue, dyspnea, pain in the lower limbs. Subjects with possible contraindications to the execution of an aerobic training (belonging to risk classes according to World Health Organization (WHO) classification and to the American College of Sports Medicine) and the execution of the MR (e.g., claustrophobia, pacemakers, pregnancy, etc.) will not be enrolled in the study. The occurrence of side effects will be recorded at each clinical visit or treatment session.

   Treatment For each subject, the treatment will lasts 8 weeks. Each treatment will consists of 35 minutes of training, administered 3 times per week. Both experimental and control treatment will be performed by two experienced physiotherapists (different from those involved in clinical and functional evaluations). Subjects of the experimental groups (both patients and HC) will carry out an aerobic training of moderate intensity (fixed time and variable intensity) on a treadmill. The training will be set individually via direct method: during the first session, the subject will be trained at an intensity that gets the heart rate (HR) corresponding to 46-63% of VO2 peak measured during the exercise test; in subsequent sessions the intensity will increase to maintain the same HR, which will be always monitored. The intensity workout identified will be maintained for 30 minutes each session, preceded and followed by a few minutes of warm-up and cool-down. Control groups of both patients and HC will follow a conventional non-aerobic physiotherapy training, structured in: 15 minutes of passive mobilization of upper and lower limbs and spine, 5 minutes of stretching of the upper and the lower limbs and 10 minutes of balance training.

   Duration The treatment period for each patient is 8 weeks. Follow-up visits will occur at 3 months after the end of treatment.

   MRI analysis All anonymized MRI data will be saved on a Linux workstation and coded with letters (A,B,C,D) according to the study group (to preserve blindness). All image post-processing will be performed by an experienced observer unaware of subjects identity and type of treatment.

   At baseline, T2 lesion volumes (LV) will be measured. New T2-visible lesions at follow up will be counted.

   On 3D T1 images, the normalized brain volume, as well as the normalized WM and GM volumes will be quantified using the cross-sectional version of the software Structural Imaging Evaluation of Normalized Atrophy (SIENAx). Longitudinal changes of brain volumes will be evaluated with the longitudinal version of the software Structural Imaging Evaluation of Normalized Atrophy (SIENA).

   Definition of the patterns of GM volume changes Voxel-based Morphometry (VBM) with Diffeomorphic Image Registration Algorithm (DARTEL) method will be applied to determine the differences of GM volumes between different subgroups of patients and controls at baseline.

   Tensor-based Morphometry (TBM) will be applied to map the longitudinal regional variations of GM volume at T1 and T2.

   Tract-based Spatial Statistics (TBSS) will be used to define the patterns of the microstructural WM abnormalities at baseline and their variations during the follow up.

   Analysis of fMRI data Active and RS fMRI data will be pre-processed using SPM12. Activations during the Stroop task will be estimated using SPM12. An independent Component Analysis (ICA) will be used to decompose RS fMRI data into spatially independent maps and time courses, using the Group ICA Of fMRI Toolbox (GIFT) software.

   Statistical analysis Demographic, clinical, functional and neuropsychological variables, as well as MRI measures at baseline will be compared using Chi-Square, t-test or ANCOVA models as appropriate. The condition of a normal distribution will be verified using the Kolmogorov-Smirnov and Shapiro-Wilk, as well as with the visual assessment of the estimated non-parametric Kernel density and Q-plot.

   To assess changes over time of clinical measures, functional and Z-score average of RS fluctuations, longitudinal linear models will be applied using a statistical design that takes into account the repeated measures in the context of a bivariate model. The correlations in each patient will be quantified with a matrix of correlations unstructured.

   The dependent variable will be the vector of the assessment from all participants at each time point (before and after treatment).

   Considering the two groups of patients together, the effects of different treatment will be evaluated considering the cross-interaction "treatment x time" in the linear model. A p value <0.05 will be considered statistically significant.

   Statistical analyses of the VBM, the TBM and the fMRI active task will be performed using the SPM12 software (whole brain analysis, p <0.05, family-wise error [FWE], corrected for multiple comparisons).

   Voxelwise differences of mean diffusivity and fractional anisotropy values between treatment and control groups at baseline, and their within-group changes at follow up will be tested, using a permutation method ("Randomize" program within FSL) and two-sample and paired t tests, as appropriate (p<0.05 FWE).

   Linear regression analysis (using SPM12) will be used to assess the correlations between fMRI activations and clinical and neuropsychological data.

   Sample size calculation Given the exploratory nature of the project, the sample size of the study has been calculated also taking into account its feasibility. The power's study showed that, for two continuous variables, with n=40 subjects and a type I error alpha= 0.05, we will able to detect a significant Pearson correlation at least equal to 0.48 with a power of 0.90 and a standardized difference between balanced groups equal to 0.8 with a power of 0.90. Furthermore, the sample size planned in this project is usually considered adequate for the performance of a fMRI analysis.

   Ethical and regulatory considerations This clinical study will be conducted in accordance with the principles laid down by the 18th World Medical Assembly (Helsinki, 1964) and all applicable amendments laid down by the World Medical Assemblies, and the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) guidelines for Good Clinical Practice.

   This clinical study will be conducted in compliance with all international laws and regulations, and national laws and regulations of the country(ies) in which the clinical trial is performed, as well as any applicable guidelines.

ELIGIBILITY:
Inclusion criteria (All)

* Age between 18 and 65 years;
* Native italian language speaking;
* Right-handed;
* No particular motor skills;
* No additional neurologic, psychiatric, orthopaedic or rheumatologic diseases;
* Normal or corrected-to-normal vision;
* No contraindications to MRI;
* Ability to understand the purpose of the study and provide signed informed consent.

For MS patients, the following additional inclusion criteria will be applied:

* Patients with a diagnosis of MS, regardless of sex, duration and course of the disease;
* EDSS score ranging from 0 to 6.0 (included);
* Stable treatment for MS from at least 1 month prior to study enrolment;
* Relapse- and steroid-free from at least 3 months before screening visit;
* An indication to perform a physiotherapy treatment by the treating physician.

Exclusion Criteria:

* Persons who perform regularly a structured training;
* Patients who performed a physiotherapy treatment for at least 3 months;
* Concomitant therapy with antidepressant, baclofen, psychoactive, and steroids drugs as well as symptomatic treatment for fatigue;
* History of alcohol or substance abuse;
* Pregnancy or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-06-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Longitudinal changes of brain GM volumes following aerobic training or conventional motor training | 2 months
  Tensor-Based Morphometry will be applied on 3D T1-weighted sequence to evaluate regional GM volume changes that will be reported as t values, ranging from 0 (no statistically significant changes) to infinity (highly statistically significant changes).
Longitudinal changes of WM microstructural abnormalities following aerobic training or conventional motor training | 2 months
  Tract-based Spatial Statistics will be applied on diffusion-tensor MRI sequence to evaluate longitudinal changes of fractional anisotropy (a dimensionless quantity ranging from 0 [more severe damage] to 1 [less severe damage]), mean diffusivity (expressed in [(mm^2)/s]×10^-3 and ranging from 0 [less severe damage] to infinity [more severe damage]), axial diffusivity (expressed in [(mm^2)/s]×10^-3 and ranging from 0 [less severe damage] to infinity [more severe damage]) and radial diffusivity (expressed in [(mm^2)/s]×10^-3 and ranging from 0 [less severe damage] to infinity [more severe damage]). Longitudinal WM microstructural changes will be reported as t values, ranging from 0 (no statistically significant changes) to infinity (highly statistically significant changes).
Resting State Functional Connectivity MRI changes following aerobic training or conventional motor training | 2 months
  Group independent component analysis Of fMRI Toolbox (GIFT) software will be applied to evaluate the modifications of resting state functional connectivity. This will be reported as z-scores, ranging from minus infinity (reduced connectivity) to infinity (increased connectivity).
  Longitudinal changes in resting state functional connectivity will be obtained subtracting baseline z-score to z-score at follow-up. A positive score means increased connectivity, a negative score, a decreased connectivity.
Functional MRI changes following aerobic training or conventional motor training | 2 months
  Statistical Parametric Mapping 12 will be applied to functional MRI sequence acquired during the Stroop task to evaluate the modifications of functional activations during this cognitive task. They will be reported as t values, ranging from 0 (no statistically significant changes) to infinity (highly statistically significant changes).
Effects of aerobic training compared to conventional motor training on global clinical disability | 2 months
  Rating of Expanded Disability Status Scale (EDSS) score changes: EDSS is a scale ranging from 0 (no disability) to 10 (death due to multiple sclerosis). Longitudinal changes will be obtained subtracting baseline EDSS to EDSS at follow-up. A positive score means disability worsening, a negative score, an improvement in disability.
Effects of aerobic training compared to conventional motor training on clinical disability | 2 months
  Rating of Multiple Sclerosis Functional Composite (MSFC) score changes: the MSFC a composite score ranging from minus infinity (worse performances) to infinity (better performances) obtained from the sum of the z-scores derived from 1) Paced Auditory Serial Addition Test (PASAT) to evaluate cognitive functions, 2) timed 25-foot walk test to evaluate walking speed, and 3) nine-hole peg test to evaluate arm and hand dexterity. Longitudinal changes will be obtained subtracting baseline MSFC to MSFC at follow-up. A positive score means disability improvement, a negative score, a worsening in disability.
Effects of aerobic training compared to conventional motor training on behavioural measures | 2 months
  Rating of functional Independent measurement (FIM) scale changes: the FIM scale is an 18-item of physical, psychological and social functions, ranging from 18 (worse disability) to 126 (total autonomy) and obtained from the sum of 18 items, each of them ranging from 1 to 7. Longitudinal changes will be obtained subtracting baseline FIM to FIM at follow-up. A positive score means behavioural improvements, a negative score, a worsening in behavioural functions.
Effects of aerobic training compared to conventional motor training on spasticity | 2 months
  Rating of Modified Ashworth Scale changes: the Modified Ashworth Scale is a 6-point scale, ranging from 0 to 4, where lower scores represent normal muscle tone and higher scores represent spasticity or increased resistance to passive movement.
  Longitudinal changes will be obtained subtracting baseline Modified Ashworth scale to Modified Ashworth scale at follow-up. A positive score means spasticity worsening, a negative score, an improvement in spasticity.
Effects of aerobic training compared to conventional motor training on walking ability | 2 months
  Assessment of Six minutes walking test changes: this is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. It is expressed in meters and ranges from 0 (worse performance) to infinity (better performance).
  Longitudinal changes will be obtained subtracting baseline distance to distance walked at follow-up. A positive score means walking improvement, a negative score, a worsening of walking ability.
Effects of aerobic training compared to conventional motor training on person's mobility | 2 months
  Assessment of Time up-and-go test changes: this is test assessing both static and dynamic balance. It uses the time (expressed in seconds) that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. It ranges from 0 (better performance) to infinity (worse performance).
  Longitudinal changes will be obtained subtracting baseline seconds to seconds needed at follow-up. A positive score means performance worsening, a negative score, an improvement in the performance.

SECONDARY OUTCOMES:
Effects of aerobic training compared to conventional motor training on cognitive functions | 2 months
  Longitudinal changes of the performances at the Brief Repeatable Battery of Neuropsychological Tests and Digit Span (forward and backward): Longitudinal changes will be obtained subtracting baseline z-scores to z-scores at follow-up. A positive score means cognitive improvement, a negative score, a worsening of cognitive performance.
Effects of aerobic training compared to conventional motor training on fatigue | 2 months
  Assessment of Modified Fatigue Impact Scale (MFIS) changes: The MFIS score is a composite score that can range from 0 (no fatigue) to 84 (highest fatigue) and that is computed by adding sub-scores from physical, cognitive, and psychosocial subscales. Longitudinal changes will be obtained subtracting baseline MFIS to MFIS at follow-up. A positive score means fatigue worsening, a negative score, an improvement in fatigue.
Effects of aerobic training compared to conventional motor training on depression | 2 months
  Assessment of Beck Depression Inventory II (BDI-II) changes: the BDI-II is a 21-question multiple-choice self-report inventory ranging from 0 (no depression to 63 severe depression). The MFIS score is a composite score that can range from 0 (no fatigue) to 84 (highest fatigue) and that is computed by adding sub-scores from physical, cognitive, and psychosocial subscales. Longitudinal changes will be obtained subtracting baseline BDI-II score to BDI-II score at follow-up. A positive score means depression, a negative score, an improvement in depression.
Effects of aerobic training compared to conventional motor training on quality of life | 2 months
  Assessment of Multiple Sclerosis Quality of Life Scale (MSQOL-54) changes: the MSQOL-54 is a 54-item scale generated from 12 subscales and two additional single-item measures and ranging from 0 (worse quality of life) to 100 (better quality of life). Longitudinal changes will be obtained subtracting baseline MSQOL-54 to MSQOL-54 at follow-up. A positive score means quality of life improvement, a negative score, a worsening of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Filippi, MD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
The dataset including all the data obtained from this study will be available from the Principal Investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The dataset including all the data obtained from this study will be available 6 months after the publication of the results.
Access Criteria: The dataset including all the data obtained from this study will be available from the Principal Investigator upon reasonable request.

REFERENCES:
- [Background] Motl RW, Pilutti LA. The benefits of exercise training in multiple sclerosis. Nat Rev Neurol. 2012 Sep;8(9):487-97. doi: 10.1038/nrneurol.2012.136. Epub 2012 Jul 24. PMID 22825702
- [Background] Prakash RS, Snook EM, Motl RW, Kramer AF. Aerobic fitness is associated with gray matter volume and white matter integrity in multiple sclerosis. Brain Res. 2010 Jun 23;1341:41-51. doi: 10.1016/j.brainres.2009.06.063. Epub 2009 Jun 25. PMID 19560443
- [Background] Ashburner J. A fast diffeomorphic image registration algorithm. Neuroimage. 2007 Oct 15;38(1):95-113. doi: 10.1016/j.neuroimage.2007.07.007. Epub 2007 Jul 18. PMID 17761438
- [Background] Leow AD, Klunder AD, Jack CR Jr, Toga AW, Dale AM, Bernstein MA, Britson PJ, Gunter JL, Ward CP, Whitwell JL, Borowski BJ, Fleisher AS, Fox NC, Harvey D, Kornak J, Schuff N, Studholme C, Alexander GE, Weiner MW, Thompson PM; ADNI Preparatory Phase Study. Longitudinal stability of MRI for mapping brain change using tensor-based morphometry. Neuroimage. 2006 Jun;31(2):627-40. doi: 10.1016/j.neuroimage.2005.12.013. Epub 2006 Feb 15. PMID 16480900
- [Background] Smith SM, Jenkinson M, Johansen-Berg H, Rueckert D, Nichols TE, Mackay CE, Watkins KE, Ciccarelli O, Cader MZ, Matthews PM, Behrens TE. Tract-based spatial statistics: voxelwise analysis of multi-subject diffusion data. Neuroimage. 2006 Jul 15;31(4):1487-505. doi: 10.1016/j.neuroimage.2006.02.024. Epub 2006 Apr 19. PMID 16624579
- [Background] Calhoun VD, Adali T, Pearlson GD, Pekar JJ. A method for making group inferences from functional MRI data using independent component analysis. Hum Brain Mapp. 2001 Nov;14(3):140-51. doi: 10.1002/hbm.1048. PMID 11559959
- [Background] Nichols TE, Holmes AP. Nonparametric permutation tests for functional neuroimaging: a primer with examples. Hum Brain Mapp. 2002 Jan;15(1):1-25. doi: 10.1002/hbm.1058. PMID 11747097
- [Background] Hayasaka S, Peiffer AM, Hugenschmidt CE, Laurienti PJ. Power and sample size calculation for neuroimaging studies by non-central random field theory. Neuroimage. 2007 Sep 1;37(3):721-30. doi: 10.1016/j.neuroimage.2007.06.009. Epub 2007 Jun 18. PMID 17658273
- [Background] Friston KJ, Holmes AP, Price CJ, Buchel C, Worsley KJ. Multisubject fMRI studies and conjunction analyses. Neuroimage. 1999 Oct;10(4):385-96. doi: 10.1006/nimg.1999.0484. PMID 10493897